CLINICAL TRIAL: NCT03315910
Title: Implementing Tobacco Treatment in Low Dose CT Lung Cancer Screening Sites
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-500
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation
Keywords: Tobacco Treatment; Lung CT; Cancer Screening; 17-500
MeSH Terms: conditions — Smoking Cessation | interventions — Motivational Interviewing; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: The investigators have chosen to conduct a full factorial experimental design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Motivational Interviewing( MI) (Yes vs. No) (Experimental): Participants will receive two motivational informed cessation sessions; the first delivered face to faceor via telephone by the SC during the patient's initial lung cancer screening visit or during the shared decision making discussion or within about 1 week following their screening visit, and the second session delivered by telephone by the SC approximately 4 to 8 weeks after the first MI session.
  Interventions: Behavioral: Motivational Interviewing (MI); Other: saliva sample
- Nicotine Replacement Therapy (NRT) Patch (Yes vs. No) (Experimental): Participants will receive 6 weeks of NRT patch with dosing dependent upon reported baseline cigarettes per day and written instructions to use the patch daily starting on date they mutually agreed upon with their site coordinator. Participants who smoke fewer than 10 cigarettes per day will receive 4-weeks of the 14mg patch (2 boxes), and 2-weeks of the 7mg patch (1 box). Those who smoke 10 or more cigarettes per day will receive 4-weeks of the 21mg patch (2 boxes) and 2-weeks of the 14mg patch (1 box). Participants will receive their study medications from their site coordinator on the day of their screening appointment or via mail from Arrowhead Promotion & Fulfillment.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Other: saliva sample
- NRT Lozenge (Yes vs. No) (Experimental): Participants will receive will receive 6 packs of NRT 2mg lozenge and written instructions to use the lozenge PRN to help manage acute nicotine withdrawal. Participants will be instructed to use the NRT lozenges no more than every 1-2 hours as needed. Participants will receive their study medications from their site coordinator on the day of their screening appointment or via mail from Arrowhead Promotion & Fulfillment.
  Interventions: Drug: Nicotine Lozenge; Other: saliva sample
- Message Framing (Gain vs. Loss) (Experimental): Overall, a robust body of health communication literature demonstrates that gain-framed messages may be more effective than loss-framed or non-framed (neutral) messages for encouraging smoking cessation. In other words, quitting messages that promote smoking cessation are more persuasive if they emphasize the benefits of quitting (gain-framed) rather than the risks (loss-framed) of persistent smoking (25, 26). Included with the written communication of their LDCT-LCS results, participants will receive a printed individualized quitting message that emphasizes either the benefits of quitting (gain-framed) or the risks of continuing to smoke (loss-framed).
  Interventions: Behavioral: Message Framing; Other: saliva sample

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — two counseling sessions
  Arms: Motivational Interviewing( MI) (Yes vs. No)
Drug: Nicotine Replacement Therapy (NRT) — receive 6 weeks of NRT patch with dosing dependent upon reported baseline cigarettes per day
  Arms: Nicotine Replacement Therapy (NRT) Patch (Yes vs. No)
Drug: Nicotine Lozenge — 6 packs of NRT 2mg lozenge
  Arms: NRT Lozenge (Yes vs. No)
Behavioral: Message Framing — health communication literature and quitting messages
  Arms: Message Framing (Gain vs. Loss)
Other: saliva sample — saliva samples from those reporting abstinence and analyze samples

SUMMARY:
This study is to help determine the most effective type or combination of treatments to offer patients seeking lung cancer screening who are smokers to help them reduce the number of cigarettes they smoke, or quit smoking. The investigators long term goal is to increase the benefits of lung cancer screening by providing a blue print of best practices for screening sites to deliver tobacco treatment to their patients who are smokers, in a way that does not add burden to screening site staff and increases the chances of patients quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

Site Eligibility (as per SC self-report)

& Must be designated as an American College of Radiology (ACR) designated lung cancer screening site

* Reports at least one year of lung cancer screening experience
* Reports conducting at least 20 new initial screenings per month Site Coordinator (SC) Eligibility (as per SC self-report)
* Employed as a full-time Site Coordinator at participating lung cancer screening site Patient Eligibility (as per self-report)
* Between the ages of 50-80 years old
* Seeking baseline or annual follow-up LDCT lung cancer screening
* Have at least a 20 pack-year history of smoking
* Currently a smoker, defined as self-reported cigarette smoking (some days, every day) within the past 30 days.
* Must be reachable by telephone
* Must be English or Spanish speaking due to the study materials being available in only these languages and limited available resources for translation.

Exclusion Criteria:

Patient (as per self-report)

* NRT is medically contraindicated (e.g., recent heart attack within the last 2 weeks or, unstable/worsening angina).
* Smokers who are receiving other tobacco treatment services or have used cessation medications (NRT, bupropion, varenicline) within the past month.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
number of patients who are tobacco abstinence | 6 months following study enrollment
  biochemical verification of smoking abstinence will be conducted Consistent with Intent to Treat, unless self reported smoking abstinence is biochemically verified, (<3 ng/ml for mailed salivary cotinine assay) for participants who fail to return the saliva sample, the cessation outcome will be considered non-abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (18):
- United States (18):
  - University of Southern California (Data Collection Only), Los Angeles, California
  - John Muir Health, Walnut Creek, California
  - WellStar Health System, La Grange, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Riverside Healthcare, Kankakee, Illinois
  - St. Mary Medical Center, Community Healthcare System, Crown Point, Indiana
  - MercyOne Des Moines Medical Center (Data Collection Only), Des Moines, Iowa
  - Maine Medical Center Cancer Institute, Scarborough, Maine
  - Henry Ford Hospital (Data collection only), Detroit, Michigan
  - Munson Healthcare, Traverse City, Michigan
  - NYU Winthrop Hospital, Mineola, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center (Data Collection Only), The Bronx, New York
  - Carolinas Healthcare System Blue Ridge, Morganton, North Carolina
  - Fairfield Medical Center, Lancaster, Ohio
  - Legacy Health, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Ostroff JS, Shelley DR, Chichester LA, King JC, Li Y, Schofield E, Ciupek A, Criswell A, Acharya R, Banerjee SC, Elkin EB, Lynch K, Weiner BJ, Orlow I, Martin CM, Chan SV, Frederico V, Camille P, Holland S, Kenney J. Study protocol of a multiphase optimization strategy trial (MOST) for delivery of smoking cessation treatment in lung cancer screening settings. Trials. 2022 Aug 17;23(1):664. doi: 10.1186/s13063-022-06568-3. PMID 35978334
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm